CLINICAL TRIAL: NCT04156048
Title: A Prospective, Epidemiologic and Multicentre Trial to Determine the Cardiovascular Risk, New Cardiovascular Events and the Cardiovascular Diseases in HIV-infected Patients: 12,5 Year Follow up
Brief Title: HIV&HEART Aging Study (12,5 Year Follow up)
Acronym: HIV&HEART
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Stefan Esser M.D., PD Dr. med. Stefan Esser, University Hospital, Essen
Other Study IDs: 12-4970-BO B
Record Dates: First submitted 2019-10-21; First posted 2019-11-07 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections; Coronary Disease; Myocardial Infarction; HIV Encephalopathy; Aging; Heart Failure
Keywords: HIV; AIDS; Antiretroviral therapy; Aging; Heart failure; coronary heart disease; myocardial infarction; HIV-associated neurocognitive disorders
MeSH Terms: conditions — HIV Infections; Coronary Disease; Myocardial Infarction; AIDS Dementia Complex; Heart Failure; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stored blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The HIV/HEART Aging study (HIVH) is an ongoing, prospective, multicentre trial that was conducted to assess the incidence, the prevalence and the clinical course of cardiovascular diseases (CVD) in HIV-infected patients. The study population includes outpatients from specialized HIV-care units of the German Ruhr region, who were at least 18 years of age, were known to have a HIV-infection and exhibited a stable disease status within 4 weeks before inclusion into the trial. From March 2004 (Pilot phase) to October 2019 (12,5 year Follow-up) 1806 HIV+ patients were recruited in a consecutive manner. The standardised examinations included a targeted assessment of medical history and physical examination. Blood was drawn for comprehensive laboratory tests including HIV specific parameters (CD4 cell count, HIV-1 RNA levels) and cardiovascular items (lipid concentrations, BNP values and renal parameters). Furthermore, non-invasive tests were performed during the initial visit, including additional heart rate and blood pressure measurements, electrocardiogram (ECGs) and transthoracic echocardiography (TTE). Examinations were completed in accordance with previously defined standard operating procedures. CVD were defined as coronary, cerebrovascular, peripheral arterial disease, heart failure or cardiac vitium.

DETAILED DESCRIPTION:
A comprehensive detailed description of the study procedures had been previously published (European Journal of medical research 2007;12:243-248).

Comprehensive non invasive cardiovascular examination

* Anamnesis
* File recherche,Physical examination
* Documentation of the cardiovascular and antiretroviral medical therapy
* Electrocardiogram
* Transthoracic echocardiography
* Exercise electrocardiogram
* Exercise Montreal Cognitive Assessment test
* Exercise the Grooved Pegboard test
* Blood collection
* Questionnaire to quality of life and health economics

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Signed informed consent

Exclusion Criteria:

* Acute cardiovascular disease
* Unstable hemodynamic status in the three weeks before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population affected by HIV
Sampling Method: Probability Sample
Enrollment: 1809 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Diseases in HIV-infected Patients | Baseline up to 12,5 year follow up

SECONDARY OUTCOMES:
Impact of classic cardiovascular risk factors of coronary artery disease, comorbidities and antiretroviral therapy | Baseline up to 12,5 year follow up
Impact of new HIV-specific risk factors of coronary artery disease, comorbidities and antiretroviral therapy | Baseline up to 12,5 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Esser, PD, MD, Principal Investigator — Departement of dermatology and venerology
Locations (6):
- Germany (6):
  - Universitätsklinikum Essen, Klinik für Dermatologie, Essen, Nordrheinwestfalen
  - University Hospital of Bochum, Department of Dermatology, Bochum, North Rhine-Westphalia
  - HIV physician pratice, Duisburg, North Rhine-Westphalia
  - Institut für Medizinische Informatik, Biometrie und Epidemiologie, Essen, North Rhine-Westphalia
  - Clinical Coordinating Center Leipzig, Leipzig, Saxony
  - HIV Outpatient Department, Dortmund